CLINICAL TRIAL: NCT04927468
Title: The Management of Large-angle Strabismus in Grave's Ophthalmopathy With Supramaximal Rectus Recession
Brief Title: Supramaximal Rectus Recession for Strabismus in Grave's Ophthalmopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Principal Investigator, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: yanghs20210607
Record Dates: First submitted 2021-06-08; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Strabismus, Mechanical; Graves Ophthalmopathy
MeSH Terms: conditions — Strabismus; Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supramaximal rectus recession (Experimental): supramaximal rectus recession to treat large-angle restricted strabismus in thyroid associated ophthalmopathy
  Interventions: Procedure: supramaximal rectus recession
- normal rectus recession (Active Comparator): normal rectus recession to treat large-angle restricted strabismus in thyroid associated ophthalmopathy
  Interventions: Procedure: normal rectus recession

INTERVENTIONS:
Procedure: supramaximal rectus recession — inferior rectus recession is 10mm，medial rectus recession is 9mm,superior rectus recession is 14mm for large-angle strabismus
  Arms: supramaximal rectus recession
Procedure: normal rectus recession — inferior rectus recession is 7mm，medial rectus recession is 7mm,superior rectus recession is 7mm for large-angle strabismus
  Arms: normal rectus recession

SUMMARY:
The purpose of this study is to evaluate supramaximal rectus recession for strabismus in Grave's Ophthalmopathy

DETAILED DESCRIPTION:
To evaluate the effectiveness and complications of supramaximal rectus recession for large-angle strabismus in Grave's Ophthalmopathy

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Grave's ophthalmopathy
* angle of deviation more than 20°
* clinically and biochemically euthyroid for at least 3 months;
* a stable orthoptic examination for at least 3 months, for example no greater than five prism dioptre change in primary position and no greater than an 8° change in duction
* monocular and mainly single extraocular muscle restricted motility

Exclusion Criteria:

* Patients with suppression, previously diagnosed and/or treated strabismus not related to the thyroid
* best-corrected visual acuity (BCVA) less than 0.2 in one or both eyes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative deviations | 6 weeks
  Postoperative deviations in the primary position were measured in prism diopters
Postoperative deviations | 3 months
  Postoperative deviations in the primary position were measured in prism diopters
Postoperative deviations | 6 months
  Postoperative deviations in the primary position were measured in prism diopters

SECONDARY OUTCOMES:
binocular single vision | 6 weeks
  measure the triple visual function including simultaneous vision, fusion range and distance stereoacuity with synoptophore.
binocular single vision | 3 months
  measure the triple visual function including simultaneous vision, fusion range and distance stereoacuity with synoptophore.
binocular single vision | 6 months
  measure the triple visual function including simultaneous vision, fusion range and distance stereoacuity with synoptophore.
stereoacuity | 6 weeks
  measure near stereoacuity in downgaze position and distance stereoacuity in primary position with random-dot stereopsis.
stereoacuity | 3 months
  measure near stereoacuity in downgaze position and distance stereoacuity in primary position with random-dot stereopsis.
stereoacuity | 6 months
  measure near stereoacuity in downgaze position and distance stereoacuity in primary position with random-dot stereopsis.
ocular motility | 6 weeks
  evaluate the ocular motility with fixed visual field examination ,scaled from -4 to +4
ocular motility | 3 months
  evaluate the ocular motility with fixed visual field examination,scaled from -4 to +4
ocular motility | 6 months
  evaluate the ocular motility with fixed visual field examination,scaled from -4 to +4

IPD SHARING:
Plan to Share IPD: No